CLINICAL TRIAL: NCT05399316
Title: The Effect of the Prebiotic Fiber INulin on metaboLITE Production of the Gut Microbiota in Healthy Adults- a Randomized, Double Blind Placebo-controlled Study
Brief Title: Inulin and the Gut Microbiota in Healthy Adults
Acronym: INLITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Experimental and Clinical Research Center (Other)
Responsible Party: Principal Investigator, Victoria McParland, Principal Investigator, Experimental and Clinical Research Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: INLITE
Record Dates: First submitted 2022-05-05; First posted 2022-06-01 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Gut Microbiota Dysbiosis and Nutrition
MeSH Terms: interventions — Inulin; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants and study staff are blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inulin (Active Comparator): 15g of powdered inulin is given in a sachet. The powder is dissolved in water and consumed
  Interventions: Dietary Supplement: Inulin
- Maltodextrin (Placebo Comparator): 15g of powdered maltodextrin is given in a sachet. The powder is dissolved in water and consumed
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Inulin — Natural fiber supplement extracted from chicory
  Arms: Inulin
Dietary Supplement: Maltodextrin — Natural non-fermentable sugar
  Arms: Maltodextrin

SUMMARY:
In this study the effects of a fibre dietary supplement on the gut microbiome in healthy adults will be investigated. For this purpose, a 14-day dietary supplementation with inulin or placebo (maltodextrin) will be carried out in healthy adults. The main objective of the study is to investigate inulin-induced changes in gut bacterial composition, bacterial gene expression, bacterial metabolite production and associated immune system changes.

DETAILED DESCRIPTION:
Healthy volunteers between the age of 18 and 60 will be recruited. In the first week of the study baseline blood and stool sampleswill be collected and nutritional information recorded. The participants will then take 15g of inulin or maltodextrin twice per day for 14 consequetive days. Blood and stool samples will be collected daily during the inital phase of the intervention and again at the end of the intervention.

From the stool samples bacterial nucleic acids will be isolated and used for metagenomic and transcriptomic analysis. The blood samples will be used to analyse for markers of barriere function and for analysis of immune cells.

ELIGIBILITY:
Inclusion Criteria:

* Men and women in a 1:1 ratio
* Age 20 - 60 years
* Body Mass Index 18.5 - 34.9 kg/m2

Exclusion Criteria:

* Arterial hypertension, diabetes mellitus, known cardiovascular disease requiring treatment (e.g. coronary heart disease, stroke).
* Known end-organ damage to the brain, heart or kidneys
* Chronic kidney disease, need for dialysis
* Diseases or functional disorders that, in the opinion of the study doctor, preclude participation in the study
* Acute infections
* Malnutrition
* Antibiotics in the previous 4 weeks
* Regular consumption of probiotics or prebiotics
* Allergies
* Change in bodyweight of more than 2 kg in the previous 3 months
* Inability to uderstand the studie aims and study procedures
* Drug or alcohol abuse

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Metabolite associated bacterial gene expression | 12 months
  The change in bacterial expression of butyrate- and propionate-associated genes in stool samples compared to placebo, adjusted to baseline. The expression of butyrate- and propionate-associated genes is measured in stool samples by quantitative PCR (qPCR).

SECONDARY OUTCOMES:
serum butyrate | 12 months
  the change in butyrate measured in serum

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Wilck, MD, Principal Investigator — Charite University; Hendrik Bartolomaeus, MD, Principal Investigator — Charite University; Victoria McParland, PhD, Principal Investigator — ECRC
Locations (1):
- Experimental and Clinical Research Center, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No